CLINICAL TRIAL: NCT01257178
Title: A Single Dose Pharmacokinetics Study of LY2624803 in Subjects With Hepatic Impairment
Brief Title: A Study to Evaluate the Pharmacokinetics of LY2624803 in Subjects With Hepatic Impairment
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial was Terminated prior to subjects receiving study drug; no trial results
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12809; I2K-MC-ZZBL (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-12-07; First posted 2010-12-09 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Normal hepatic function (Experimental): 6mg, oral, once on day 1
  Interventions: Drug: LY2624803
- Mild hepatic impairment (Experimental): 6 mg, oral, once on day 1
  Interventions: Drug: LY2624803
- Moderate hepatic impairment (Experimental): 6 mg, oral, once on day 1
  Interventions: Drug: LY2624803
- Severe hepatic impairment (Experimental): 6 mg, oral, once on day 1
  Interventions: Drug: LY2624803

INTERVENTIONS:
Drug: LY2624803 — Administered orally

SUMMARY:
The purpose of this study is to evaluate the impact of hepatic dysfunction on the pharmacokinetics and safety of LY2624803 and its major metabolite, LSN2797276.

ELIGIBILITY:
Inclusion Criteria:

All Subjects

* Sexually active male and female subjects and their partners must agree to use 2 methods of contraception such as condom or occlusive cap (diaphragm or cervical/vault caps) together with spermicidal foam/gel/film/cream/suppository, from the time the subject enters the study until 3 months after the final dosing occasion, unless the male subject or partner has been sterilized (with confirmed azoospermia).
* Have a BMI between 18.5 and 35.0 kg/m2, inclusive.
* Have a body weight >50 kg.
* Have normal sitting blood pressure and heart rate compatible with their disease state, as determined by the investigator.
* Have venous access sufficient to allow blood sampling as per the protocol.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Have given written informed consent approved by Lilly and the Ethical Review Board governing the site.

Control Subjects

* Are males or females and with normal hepatic function, as determined by medical history and physical examination.
* Have clinical laboratory test results within normal reference range for the investigator site, or results with minor deviations not considered to be clinically significant by the investigator.

Hepatic Impaired Subjects

•Have stable hepatic impairment (alcoholic, posthepatitis, biliary cirrhosis, cryptogenic) classified as Child-Pugh class A, B, or C (mild, moderate, and severe impairment) who are considered acceptable for participation in the study by the investigator.

Exclusion Criteria:

All Subjects

* Are currently enrolled in, or discontinued within the last 90 days from the last dosing occasion in a clinical trial involving an investigational drug or device, or are concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.
* Have known allergies to LY2624803 or related compounds.
* Have previously discontinued from this study or any other study investigating LY2624803.
* Have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk associated with participating in the study.
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening.
* Show evidence of human immunodeficiency virus (HIV) and/or positive HIV antibodies.
* Have donated blood of more than 500 mL within the last 3 months prior to the screening visit.
* Use drugs or herbal remedies that are known inhibitors or inducers of CYP3A4 or inhibitors of CYP2D6 enzyme pathways, unless in the opinion of the sponsor and investigator the medication will not compromise safety.
* Are liver transplant subjects or have taken immunosuppressants following any organ transplant.
* Have shown signs of variceal bleeding during the last 2 weeks prior to screening.
* Show evidence of irritable bowel syndrome or chronic diarrhea.
* Have an average weekly alcohol intake that exceeds 28 units per week (males) and 21 units per week (females), and are subjects unwilling to stop alcohol consumption for the duration of the study (1 unit = 12 oz or 360 mL of beer; 5 oz or 150 mL of wine; 1.5 oz or 45 mL of distilled spirits).
* Are unable to swallow whole capsules.
* Are on total parenteral nutrition (TPN).
* Take anticoagulants for therapeutic use.
* Have a history of breast cancer.
* Exhibit any other condition, which, in the opinion of the investigator would preclude participation in the study.

Control Subjects

* Have any medically significant history of neurologic disease, cancer, or cardiac, respiratory, metabolic, hepatic, renal, gastrointestinal (except appendectomy), dermatological, venereal, hematological disorder or disease.
* Have creatinine clearance (CrCl) <80 mL/min, as calculated by Cockcroft-Gault equation.
* Show evidence of significant active neuropsychiatric disease in the opinion of the investigator.
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen (HBsAg).
* Show evidence of hepatitis C and/or positive hepatitis C antibody.

Mild Hepatic Impaired Subjects (Child-Pugh A)

* Show evidence of any significant active disease other than that responsible for or associated with hepatic impairment.
* Show evidence of active renal disease with creatinine clearance <70 mL/min as calculated by Cockcroft-Gault equation.
* Have severe ascites.

Moderate and Severe Hepatic Impaired Subjects (Child-Pugh B and C)

* Show evidence of any significant active disease other than that responsible for or associated with moderate or severe hepatic impairment.
* Show evidence of hepatorenal syndrome as shown by creatinine clearance <50 mL/min, as calculated by the Cockcroft-Gault equation.
* Have shown signs of spontaneous bacterial peritonitis within 6 months prior to dosing.
* Have severe hyponatremia.
* Have hepatic encephalopathy (grade 2 to 4 encephalopathy).
* Show signs of hepatocellular carcinoma.
* Have a portal shunt.
* Show, in the opinion of the investigator, evidence of significant active neuropsychiatric disease other than grade 1 hepatic encephalopathy.
* Have severe ascites.
* Have hemoglobin concentrations <9.0 g/dL.
* Have a platelet count of <50 x 109 cells/L, unless, after consultation with the sponsor, they are considered as acceptable for participation in the study.
* Have total serum bilirubin concentrations >15 mg/dL (>257 µmol/L).
* Take medications known to interfere with hepatic metabolism (for example barbiturates, phenothiazines) or known to alter other major organ systems.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
LY2624803 and the metabolite LSN2797276 Area under the Curve from time 0 to infinity [AUC(0-∞)] | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, Maximum Concentration (Cmax) | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, Time to maximum plasma concentration(tmax) | Predose through 120 hours post dose

SECONDARY OUTCOMES:
LY2624803 and the metabolite LSN2797276, Elimination half live (t1/2) | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, AUC to the last quantifiable sample [AUC(0-tlast)] | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, Apparent clearance (CL/F) | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, Apparent volume of distribution (V/F) | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, Parent to metabolite ratios (MR) of Cmax | Predose through 120 hours post dose
LY2624803 and the metabolite LSN2797276, Parent to metabolite ratios (MR) of AUC | Predose through 120 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (4):
- Germany (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mitte
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., München
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen, Hungary
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia